CLINICAL TRIAL: NCT05294029
Title: Neuro-Orthopaedic Disorders During Aging in Patients With Neuromotor Disability
Acronym: NO-AGING
Status: Recruiting | Type: Observational
Sponsor: Institut de Sante Parasport Connecte Synergies (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-002
Record Dates: First submitted 2022-01-05; First posted 2022-03-24 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Disability or Chronic Disease Leading to Disablement
Keywords: Neuromotor Disability, Neuro-Orthopaedics
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects with neuromotor disability
  Interventions: Other: standard of care for patients with neuromotor disability

INTERVENTIONS:
Other: standard of care for patients with neuromotor disability — clinical examination, radiological, biological and physiological examinations.

SUMMARY:
People with neuromotor disability (i.e. following an inborn or acquired spinal cord, cerebral or peripheral neurological lesion) are at risk of worsening their neuro-orthopaedic disorders during aging, including fracture risk. Nevertheless, at the present time, the natural evolution of their neuro-orthopedic disorders and the long-term functional impact of their medical and surgical treatments is unknown.

The aim of this study is to describe neuro-orthopedic disorders during aging of patients with neuromotor disability, their functional repercussions, their comorbidities and the therapeutic strategies used.

DETAILED DESCRIPTION:
This is an ambispective, monocentric, cohort study of subjects with neuromotor disability followed in a Physical Medicine and Rehabilitation Department.

All consecutive eligible inpatient and outpatient subjects treated in the Neuro Orthopaedic Unit (UPOH) of the Physical Medicine and Rehabilitation Department of our university hospital will be included.

Data will be collected from the patients' medical records, in particular data related to their clinical, radiological, biological and physiological examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old ;
* Treated in the Neuro Orthopaedic Unit (UPOH) of the Physical Medicine and Rehabilitation Department of our university hospital ;
* Having a neuromotor disability ;
* No opposition to be enrolled in the study from the patient, or from a legally authorized close relative if the patient's state of health does not allow it ;
* Affiliation to a social security scheme.

Exclusion Criteria:

* Under court protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with neuromotor disability
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2032-02-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of mobility during aging | Through study completion, an average of 1 year
  Walking range

SECONDARY OUTCOMES:
Prevalence of falls and fractures | Through study completion, an average of 1 year
  Number and description of falls and fractures
Characteristics of infiltrative procedures and surgeries | Through study completion, an average of 1 year
  Number and description of infiltrative procedures and surgeries
Changes of devices (orthoses and prostheses) and technical aids used during aging | Through study completion, an average of 1 year
  Number and description of devices (orthoses and prostheses) and technical aids
Changes of physical activity, as well as barriers and facilitators to physical activity, during aging | Through study completion, an average of 1 year
  Questionnaires assessing physical activity levels (ex: PASPID) and barriers and facilitators to physical activity (ex: BPAQ)
Evolution of comorbidities during aging | Through study completion, an average of 1 year
  Prevalence of comorbidities (e.g. obesity, diabetes, hypertension, sleep apnea, ...)
Medication | Through study completion, an average of 1 year
  Medication list
Prevalence of pressure sores | Through study completion, an average of 1 year
  Number and description of pressure sores

CONTACTS AND LOCATIONS:
Overall Officials: François Genêt, MD-PhD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France; Vincent T Carpentier, MD-MSc, Study Director — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France
Locations (1):
- Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, Garches, France

IPD SHARING:
Plan to Share IPD: No